CLINICAL TRIAL: NCT06017076
Title: Effect of Preoperative Oral Energy Drinks Compared to Warming Matress on Body Temperature During Combined Spinal-epidural Anesthesia for Elective Cesarean Delivery: a Randomised Non-inferiority Trial.
Brief Title: Effect of Preoperative Oral Energy Drinks Compared to Warming Matress on Body Temperature During Combined Spinal-epidural Anesthesia for Elective Cesarean Delivery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Feng, MD, Head of anesthesiology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SFY2023-MZ8-3
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2023-08

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Energy Drinks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- warming matress group (Placebo Comparator): From the end of anesthesia, warming matriss at 40 ℃ was used for insulation until the end of surgery.
  Interventions: Device: Warming matress
- oral functional drinks group (Experimental): Patients drank energy drinks (Red Bull®) 250ml about 2-2.5 hours before operation.
  Interventions: Other: Oral energy drinks

INTERVENTIONS:
Other: Oral energy drinks — Patients drank energy drinks (Red Bull®) 250ml about 2-2.5 hours before operation.
  Arms: oral functional drinks group
Device: Warming matress — From the end of anesthesia, warming matriss at 40 ℃ was used to keep warm until the end of surgery.
  Arms: warming matress group

SUMMARY:
It is not known which is better for intraoperative temperature protection, warming matress or preoperative oral functional drinks in elective cesarean section. We plan to conduct a non inferiority randomized trial to clarify this problem.

ELIGIBILITY:
Inclusion Criteria:

* Women pregnant with a single fetus;
* American Society of Anesthesiologists (ASA) physical status II;
* Willingness to undergo elective cesarean delivery under combined spinal-epidural anesthesia;
* A body mass index (BMI) < 35 kg·m-2;
* A gestational age of 38-40 weeks.

Exclusion Criteria:

* Contraindications for combined spinal-epidural anesthesia;
* A diagnosis of delayed gastric emptying, hyperemesis gravidarum until late pregnancy, or consumption of drugs that affect gastrointestinal motility within 3 days before surgery;
* Preoperative body temperature >38°C or <36°C or the use of drugs that affect body temperature;
* Pregnancy combined with diabetes, hypertension, or metabolic disorders (eg, hypothyroidism or hyperthyroidism);
* Ear diseases (eg, otitis media, tympanic membrane perforation, etc) affecting measurement of ear temperature;
* Intraoperative malfunction of the warming blanket;
* Patients who were simultaneously undergoing other operations (eg, removal of uterine fibroids and ovarian cysts) or had a surgical time >1.5 hours;
* Patients with blood transfusion or autologous blood transfusion intraoperatively;
* Patients who did not receive the anesthetic specified in the protocol;
* Patients who failed to drink 125ml energy drinks before surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2023-09-03 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Core temperature change | Before the operation, and every 10 minutes during the operation until the end of the operation.
  The minimum value of intraoperative ear temperature minus the preoperative baseline ear temperature.

SECONDARY OUTCOMES:
Skin temperature changes | Before the operation, and every 10 minutes during the operation until the end of the operation.
  The minimum value of intraoperative skin temperature minus the preoperative baseline skin temperature.
hypotension | Intraoperative
  Number of Participants with systolic blood pressure reduction >20% baseline value or systolic blood pressure <90 mm Hg before delivery
The incidence of nausea in pregnant women | Intraoperative
  Anesthesiologist observes combined patient dictation.
Umbilical artery blood base excess | 30sec after delivery
  base excess of fetal umbilical artery blood
The incidence of vomiting in pregnant women | Intraoperative
  Anesthesiologist observes combined patient dictation
The incidence of shivering in pregnant women | Intraoperative
  Anesthesiologist observes combined patient dictation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Peking University People's Hospital, 11 Xizhimen South Street, Xicheng District, Beijing, People's Republic of China, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes